CLINICAL TRIAL: NCT01169922
Title: HIV Prevention With Adolescents: Neurocognitive Deficits and Treatment Response
Acronym: SHARP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study did not begin and is being terminated from the system.
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NIAAA RO1 AA017390-01
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Risk Reduction Behavior; Sexual Behavior; Health Behavior; Drinking Behavior; Adolescent Behavior
MeSH Terms: conditions — Risk Reduction Behavior; Sexual Behavior; Health Behavior; Drinking Behavior; Adolescent Behavior | interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- SEXUAL PLUS ALCOHOL RISK REDUCTION (Experimental): Intervention contains information geared toward sexual risk reduction as well as alcohol risk reduction.
  Interventions: Behavioral: SEXUAL RISK REDUCTION + ALCOHOL RISK REDUCTION
- INFORMATION-ONLY SEXUAL RISK REDUCTION (Active Comparator): Intervention contains information geared toward sexual risk reduction only.
  Interventions: Behavioral: INFORMATION-ONLY SEXUAL RISK REDUCTION

INTERVENTIONS:
Behavioral: SEXUAL RISK REDUCTION + ALCOHOL RISK REDUCTION — 2 hour 50 minute long intervention; includes presentation of STD/HIV facts, activities/games regarding safe sex, condom demonstration, video about sexual decision making, video about alcohol/sexual decision making, alcohol-related risk-reduction motivational interview, group discussion
  Other Names: SEXUAL RISK REDUCTION + ALCOHOL RISK REDUCTION (SRRI+ETOH)
  Arms: SEXUAL PLUS ALCOHOL RISK REDUCTION
Behavioral: INFORMATION-ONLY SEXUAL RISK REDUCTION — 1 hour 30 minute long intervention; includes presentation of STD/HIV facts, video about sexually transmitted diseases, review of STD/HIV facts
  Other Names: INFORMATION-ONLY SEXUAL RISK REDUCTION (INFO-ONLY)
  Arms: INFORMATION-ONLY SEXUAL RISK REDUCTION

SUMMARY:
This research is examining how genetic and brain factors play a role in adolescents' health risk behavior as well as studying behaviors that young people engage in that may place them at risk for contracting a sexually transmitted disease like HIV/AIDS, and what kind of educational program works best to reduce these risky behaviors.

DETAILED DESCRIPTION:
A baseline assessment is conducted, including a computer questionnaire assessing personality characteristics, attitudes toward and experiences with sex, alcohol, drugs, and cigarettes, among other things. The participant also meets with a therapist to conduct a brief motivational interview at this time. A "Time-Line Follow-Back" is conducted; this notes incidences of sexual intercourse, alcohol use, marijuana use, and cigarette use in a 30-day period. An fMRI is conducted, and a saliva sample is gathered. During the second session of the study, participants are randomly assigned to either a sex and alcohol risk reduction intervention, or a sex risk reduction intervention. After the intervention, participants are contacted at 3 month intervals (3 months later, 6 months later, 9 months later, and 12 months later) to meet. At these "follow-up" meetings, another Time-Line Follow-Back is conducted, along with another computer questionnaire (again assessing attitudes toward and experiences with sex, alcohol, drugs, and cigarettes).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents age 14-18
* Involved in Juvenile Justice System OR enrolled in a private school

Exclusion Criteria:

* Currently taking anti-psychotics
* Involved in similar intervention-based study (2 similar studies being conducted simultaneously by this lab)

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Time-Line Follow-Back (TLFB) | 3-months post-intervention
  A Time-Line Follow-Back is a review of a recent 30-day period of the participant's life, wherein they note which days they engaged in any of the following activities: sexual intercourse, alcohol use, marijuana use, cigarette use. Further details are also provided, such as whether a condom was used, how many alcoholic drinks were consumed, etc.
Time-Line Follow-Back (TLFB) | 6-months post-intervention
  A Time-Line Follow-Back is a review of a recent 30-day period of the participant's life, wherein they note which days they engaged in any of the following activities: sexual intercourse, alcohol use, marijuana use, cigarette use. Further details are also provided, such as whether a condom was used, how many alcoholic drinks were consumed, etc.
Time-Line Follow-Back (TLFB) | 9-months post-intervention
  A Time-Line Follow-Back is a review of a recent 30-day period of the participant's life, wherein they note which days they engaged in any of the following activities: sexual intercourse, alcohol use, marijuana use, cigarette use. Further details are also provided, such as whether a condom was used, how many alcoholic drinks were consumed, etc.
Time-Line Follow-Back (TLFB) | 12-months post-intervention
  A Time-Line Follow-Back is a review of a recent 30-day period of the participant's life, wherein they note which days they engaged in any of the following activities: sexual intercourse, alcohol use, marijuana use, cigarette use. Further details are also provided, such as whether a condom was used, how many alcoholic drinks were consumed, etc.

SECONDARY OUTCOMES:
Computer questionnaire | 3 months post-intervention
  Questionnaire completed by participant assesses sexual activity/consequences/attitudes, alcohol use/consequences/attitudes, marijuana use/consequences/attitudes, cigarette use/consequences/attitudes within past few months
Computer questionnaire | 6 months post-intervention
  Questionnaire completed by participant assesses sexual activity/consequences/attitudes, alcohol use/consequences/attitudes, marijuana use/consequences/attitudes, cigarette use/consequences/attitudes within past few months
Computer questionnaire | 9 months post-intervention
  Questionnaire completed by participant assesses sexual activity/consequences/attitudes, alcohol use/consequences/attitudes, marijuana use/consequences/attitudes, cigarette use/consequences/attitudes within past few months
Computer questionnaire | 12 months post-intervention
  Questionnaire completed by participant assesses sexual activity/consequences/attitudes, alcohol use/consequences/attitudes, marijuana use/consequences/attitudes, cigarette use/consequences/attitudes within past few months

CONTACTS AND LOCATIONS:
Overall Officials: Angela D Bryan, PhD, Principal Investigator
Locations (4):
- United States (4):
  - Diversion Meetings (Youth Services Center), Albuquerque, New Mexico
  - Youth Reporting Center (Youth Services Center), Albuquerque, New Mexico
  - Albuquerque Academy, Albuquerque, New Mexico
  - Sandia Preparatory School, Albuquerque, New Mexico